CLINICAL TRIAL: NCT00121459
Title: The Latex Diaphragm to Prevent HIV Acquisition Among Women: A Female-Controlled, Physical Barrier of the Cervix
Brief Title: Effectiveness of the Diaphragm for HIV Prevention
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: PI left and no data or information is available.
Sponsor: University of California, San Francisco (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Ibis Reproductive Health (Other); Medical Research Council, South Africa (Other); Women's Health Global Imperative (Unknown); UZ-UCSF Collaborative Research Programme (Other); Perinatal HIV Research Unit of the University of the Witswatersrand (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H6070-22217-03; 21082
Record Dates: First submitted 2005-07-12; First posted 2005-07-21 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: HIV Infection
Keywords: Diaphragm; HIV prevention; Southern/South Africa, Zimbabwe; female-controlled methods; Replens; STI prevention; HIV Seronegativity
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Device: Ortho All-Flex diaphragm and Replens lubricant gel

SUMMARY:
The purpose of this trial is to determine whether using the diaphragm and a lubricant get can reduce women's risk of acquiring an HIV infection.

DETAILED DESCRIPTION:
This multi-site randomized, controlled trial will measure the effectiveness of the diaphragm in preventing heterosexual acquisition of HIV infection among women. This Phase III study is powered to detect effectiveness (biological efficacy combined with adherence) of 33 percent. Women in South Africa and Zimbabwe (N=4,500) at risk of contracting HIV will be invited to participate and will be followed for up to 24 months, with a total study duration of 4 years. All women will receive safer-sex counseling, free male condoms and diagnosis and treatment of sexually transmitted infections (STIs). Half of the participants will be randomly selected to receive an Ortho All-Flex latex diaphragm and Replens lubricant gel. We will assess whether women using diaphragms and lubricant gel have lower rates of HIV or STI infection than do their non-diaphragm and gel counterparts. Additionally, we will investigate the long-term acceptability of the diaphragm in this study population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 49 years old
* Sexually active (coital frequency at least four times per month on average)
* HIV negative based on testing within two weeks prior to enrollment
* Chlamydia trachomatis and Neisseria gonorrhoeae negative based on testing within 30 days prior to enrollment or if positive, completes treatment before enrollment
* Have a healthy cervix, as assessed by naked-eye speculum exam at enrollment
* Planning to live in the study area for the next 24 months
* Willing to be randomly assigned either to use or not use a latex diaphragm with lubricant gel during participation in the study, and to follow the protocol, including being tested for HIV and STIs
* Willing and able to give informed consent

Exclusion Criteria:

* Known sensitivity or allergy to latex
* History of TSS (as suggested by current labeling for diaphragm use)
* Currently pregnant, or desiring to become pregnant in the next two years
* No cervix (total hysterectomy)
* Refuses treatment for diagnosed or suspected current STI and/or reproductive tract infection requiring treatment at enrollment
* Within six weeks of any pelvic surgery or last pregnancy outcome at the time of screening and enrollment
* Presence of clinically apparent lesion(s) with epithelial disruption at enrollment (may enroll after lesion(s) has healed, if otherwise eligible)
* Injected illicit drugs in the 12 months prior to screening and enrollment
* Blood transfusion or received blood products in 3 months prior to screening and enrollment
* Unable or unwilling to insert the diaphragm correctly
* Participation in any other clinical trial (including those of a vaginal product or barrier contraceptive). Verification by comparing participant lists to other concurrently running research studies may be conducted if necessary.
* Unable to speak English, Zulu, Shona, or Sotho
* Other conditions that, in the opinion of the investigator, would constitute contraindications to participation in the study or would compromise ability to comply with the study protocol, such as a major psychiatric disorder

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2003-09

PRIMARY OUTCOMES:
HIV incidence

SECONDARY OUTCOMES:
STI incidence (CT, NG, syphilis, trichomoniasis, HSV2)
acceptability
feasibility and sustainability

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Padian, PhD, Principal Investigator — University of California, San Francisco
Locations (3):
- South Africa (2):
  - Perinatal HIV Research Unit, Soweto, Gauteng
  - Medical Research Council of South Africa, Durban, KwaZulu-Natal
- UZ-UCSF, Harare, Zimbabwe

REFERENCES:
- [Derived] Teasdale CA, Abrams EJ, Chiasson MA, Justman J, Blanchard K, Jones HE. Incidence of sexually transmitted infections during pregnancy. PLoS One. 2018 May 24;13(5):e0197696. doi: 10.1371/journal.pone.0197696. eCollection 2018. PMID 29795625
- [Derived] Abbai NS, Wand H, Ramjee G. Biological factors that place women at risk for HIV: evidence from a large-scale clinical trial in Durban. BMC Womens Health. 2016 Mar 19;16:19. doi: 10.1186/s12905-016-0295-5. PMID 26992693
- [Derived] Abbai NS, Wand H, Ramjee G. Socio-demographic and behavioural characteristics associated with HSV-2 sero-prevalence in high risk women in KwaZulu-Natal. BMC Res Notes. 2015 May 5;8:185. doi: 10.1186/s13104-015-1093-0. PMID 25940115
- [Derived] Naidoo S, Wand H, Abbai NS, Ramjee G. High prevalence and incidence of sexually transmitted infections among women living in Kwazulu-Natal, South Africa. AIDS Res Ther. 2014 Sep 15;11:31. doi: 10.1186/1742-6405-11-31. eCollection 2014. PMID 25243015
- [Derived] Ramjee G, Wand H. Geographical clustering of high risk sexual behaviors in "hot-spots" for HIV and sexually transmitted infections in Kwazulu-Natal, South Africa. AIDS Behav. 2014 Feb;18(2):317-22. doi: 10.1007/s10461-013-0578-x. PMID 23934268
- [Derived] Wand H, Ramjee G. The relationship between age of coital debut and HIV seroprevalence among women in Durban, South Africa: a cohort study. BMJ Open. 2012 Jan 5;2(1):e000285. doi: 10.1136/bmjopen-2011-000285. Print 2012. PMID 22223838
- [Derived] Blanchard K, Bostrom A, Montgomery E, van der Straten A, Lince N, de Bruyn G, Grossman D, Chipato T, Ramjee G, Padian N. Contraception use and effectiveness among women in a trial of the diaphragm for HIV prevention. Contraception. 2011 Jun;83(6):556-63. doi: 10.1016/j.contraception.2010.10.018. Epub 2011 Jan 26. PMID 21570554
- [Derived] de Bruyn G, Shiboski S, van der Straten A, Blanchard K, Chipato T, Ramjee G, Montgomery E, Padian N; MIRA Team. The effect of the vaginal diaphragm and lubricant gel on acquisition of HSV-2. Sex Transm Infect. 2011 Jun;87(4):301-5. doi: 10.1136/sti.2010.047142. Epub 2011 Mar 29. PMID 21447515
- [Derived] van der Straten A, Cheng H, Minnis AM. Change in condom and other barrier method use during and after an HIV prevention trial in Zimbabwe. J Int AIDS Soc. 2010 Oct 19;13:39. doi: 10.1186/1758-2652-13-39. PMID 20955629
- [Derived] Sawaya GF, Chirenje MZ, Magure MT, Tuveson JL, Ma Y, Shiboski SC, Da Costa MM, Palefsky JM, Moscicki AB, Mutasa RM, Chipato T, Smith-McCune KK. Effect of diaphragm and lubricant gel provision on human papillomavirus infection among women provided with condoms: a randomized controlled trial. Obstet Gynecol. 2008 Nov;112(5):990-7. doi: 10.1097/AOG.0b013e318189a8a4. PMID 18978097
- [Derived] Ramjee G, van der Straten A, Chipato T, de Bruyn G, Blanchard K, Shiboski S, Cheng H, Montgomery E, Padian N; MIRA team. The diaphragm and lubricant gel for prevention of cervical sexually transmitted infections: results of a randomized controlled trial. PLoS One. 2008;3(10):e3488. doi: 10.1371/journal.pone.0003488. Epub 2008 Oct 22. PMID 18941533
- [Derived] Padian NS, van der Straten A, Ramjee G, Chipato T, de Bruyn G, Blanchard K, Shiboski S, Montgomery ET, Fancher H, Cheng H, Rosenblum M, van der Laan M, Jewell N, McIntyre J; MIRA Team. Diaphragm and lubricant gel for prevention of HIV acquisition in southern African women: a randomised controlled trial. Lancet. 2007 Jul 21;370(9583):251-261. doi: 10.1016/S0140-6736(07)60950-7. PMID 17631387
- See also: Ibis Reproductive Health web site — http://www.ibisreproductivehealth.org
- See also: Cervical Barrier Advancement Society web site — http://www.cervicalbarriers.org
- See also: Women's Global Health Imperative — http://www.rti.org/wghi
- See also: University of Zimbabwe, UCSF — http://www.uz-ucsf.co.zw/
- See also: Medical Research Council — http://www.mrc.ac.za/hiv/hiv.htm
- See also: Perinatal HIV Research Unit of South Africa — http://www.hivsa.com/